CLINICAL TRIAL: NCT01316471
Title: Web-MAP 2: Internet Intervention for Adolescents With Chronic Pain
Brief Title: Internet Intervention for Adolescents With Chronic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Tonya Palermo, Professor, Anesthesiology and Pain Medicine, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HD062538-01A1 (NIH)
Record Dates: First submitted 2011-03-11; First posted 2011-03-16 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Chronic Pain; Abdominal Pain; Headache
Keywords: Chronic Pain; Abdominal Pain; Headache; Adolescents; Internet Interventions; Behavioral Interventions
MeSH Terms: conditions — Chronic Pain; Abdominal Pain; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Online Behavioral Intervention (Experimental): In addition to standard medical care, children and parents in the online behavioral intervention will receive access to the full web-based program including education about chronic pain, training in behavioral and cognitive coping skills, instruction in increasing activity participation, and education about pain behaviors and parental operant strategies using an engaging, interactive format on the Internet.
  Interventions: Behavioral: Online Behavioral Intervention
- Online Patient Education (Active Comparator): The Online Patient Education group will serve as an attention control condition. In addition to standard medical care, children and parents will be provided with access to a modified version of the study website that will provide information from publicly available educational websites about pediatric chronic pain management.
  Interventions: Other: Education: Online Patient Education

INTERVENTIONS:
Behavioral: Online Behavioral Intervention — The online behavioral intervention is travel-themed and participants visit 8 destinations (1 per week) designed to take 30 min each to complete. The destinations serve as an online analog for the weekly sessions used when delivering behavioral interventions face-to-face. The 8 child destinations include: 1) education about chronic pain, 2) recognizing stress and negative emotions, 3) relaxation and distraction skills, 4) school, 5) cognitive skills, 6) sleep hygiene and lifestyle, 7) staying active, and 8) relapse prevention. The eight parent destinations include: 1) education about chronic pain, 2) recognizing stress and negative emotions, 3) operant strategies I, 4) operant strategies II, 5) modeling, 6) sleep hygiene and lifestyle, 7) communication, and 8) relapse prevention.
  Other Names: Internet Intervention
  Arms: Online Behavioral Intervention
Other: Education: Online Patient Education — The purpose of the online patient education group is to control for time, attention, and computer usage. Children and parents will be provided with access to a modified version of the study website that will provide links to information from publicly available educational websites about pediatric chronic pain management. Children and parents will log onto the web program weekly at the same interval as the Online Behavioral Intervention group. Children and parents will be asked to view 3 links each week and then report a few details pertaining to the content of what they viewed.
  Other Names: Online Attention Control
  Arms: Online Patient Education

SUMMARY:
The purpose of this study is to evaluate the efficacy of a web-based (i.e., internet) behavioral program to reduce pain and improve functioning in children and adolescents with chronic pain. We hypothesize that children and adolescents in families that receive the web-based behavioral program will report reduced pain levels and improved daily functioning compared to children and their parents who receive online patient education.

DETAILED DESCRIPTION:
An estimated 15% to 30% of otherwise healthy children and adolescents suffer from recurrent or chronic pain such as headache, abdominal pain, and musculoskeletal pain. Chronic pain has a significant impact on children's mood, daily functioning, and overall quality of life. Effective behavioral interventions have been developed to increase positive coping behaviors. However, most children do not have access to these interventions due to a variety of barriers such as distance from pediatric pain treatment centers. We have developed an online behavioral intervention called Web-based Management of Adolescent Pain (Web-MAP), and our preliminary findings indicated that children in families that received this intervention experienced significant improvements in their pain level and daily functioning compared to children who did not receive the intervention (Palermo et al., 2009). The purpose of this study is to extend these findings by: 1) recruiting families from other medical centers, 2) determining whether the benefits of online behavioral intervention are maintained 6- and 12-months after the intervention has been completed, 3) evaluating additional outcomes such as parent responses to pain and child sleep quality, anxiety, depression, and health service use, 4) comparing results from online behavioral intervention to online patient education.

ELIGIBILITY:
Inclusion Criteria:

* Literate in English
* Age 11-17 years
* Pain present for at least 3 months duration
* Pain occurs at least 1 time per week and interferes with daily functioning
* Pain is not related to a chronic disease
* Receiving evaluation or treatment in a pediatric pain clinic
* Has access to a computer, the Internet, and a phone

Exclusion Criteria:

* A serious comorbid chronic condition in the patient (e.g., diabetes, arthritis, cancer).
* Non-English speaking
* More than 4 sessions of CBT for pain management in the 6 months prior to the time of screening.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 273 (Actual)
Dates: Start 2011-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Activity limitations | pre-treatment, immediately post-treatment, 6-month follow-up, 12-month follow-up
  Child report of activity limitations will be assessed using the prospective version of the Child Activity Limitations Interview (Palermo, Witherspoon, Valenzuela, & Drotar, 2004), which includes 8 activities that children identify as important in their day-to-day lives that are impacted by pain. Responses are rated on a 5-point scale (0-4) with higher scores indicating greater perceived difficulty with activities. Children will provide ratings daily for 7 days on their online diaries at each assessment period. Mean activity limitations across the reporting period is used in analyses.
Pain intensity | pre-treatment, immediately post-treatment, 6-month follow-up, 12-month follow-up
  Children will report on presence and intensity of pain daily for 7 days at each assessment period. Pain intensity will be assessed using an 11-point numerical rating scale (NRS) with anchors of 0= no pain to 10= worst pain (McGrath et al., 2008). Mean average intensity of the pain reported will serve as primary pain measure.

SECONDARY OUTCOMES:
Depression and pain-specific anxiety | pre-treatment, immediately post-treatment, 6-month follow-up, 12-month follow-up
  Children will complete the Bath Adolescent Pain Questionnaire (BAPQ), a 61-item scale that will be used to measure pain-specific emotional functioning (Eccleston et al., 2005). The BAPQ was developed specifically for children with chronic pain and has demonstrated adequate reliability and validity (Eccleston et al., 2008). For the purpose of this study, the subscales of depression and pain-specific anxiety will be used in analyses.
Treatment Satisfaction | Immediately Post-Treatment, 6-month follow-up, 12-month follow-up
  Children and parents will complete this questionnaire, which includes items that address satisfaction with the therapeutic process during the course of treatment and satisfaction with the outcome of therapy. Items are rated on a 5-point scale from 1 = strongly disagree to 5 = strongly agree.
Parental Response to Pain Behavior | pre-treatment, immediately post-treatment, 6-month follow-up, 12-month follow-up
  Children and their parents will complete the Adult Responses to Children's Symptoms (ARCS), a 29-item measure assessing parental responses to child pain behavior (Walker, Levy, & Whitehead, 2006). Respondents rate on a five-point Likert scale the frequency with which parents engage in specific behaviors in response to their child's pain.
Sleep Quality | pre-treatment, immediately post-treatment, 6-month follow-up, 12-month follow-up
  Children's perception of sleep quality will be measured by the Adolescent Sleep Wake Scale (LeBourgeois et al., 2005), a 28-item self-report scale that assesses five behavioral dimensions of teens' sleep: going to bed, falling asleep, maintaining sleep, reinitiating sleep, and returning to wakefulness. Subscale scores range from 1 to 6, with higher scores indicating better sleep quality.
Health service Use | pre-treatment, 12-month follow-up
  Parents will complete the Client Service Receipt Inventory-Pain version (Sleed et al., 2005), a measure of service use, out-of-pocket expenses, and lost work time incurred by families for the evaluation or management of the child's chronic pain. Questions pertain to hospital admissions, outpatient services, community services (e.g., tutor, lawyer), medications, lost work time, paid help, and other costs. We will compute the following variables: total number of services used, number of lost parental work days, and number of out-of-pocket expenses.
Miscarried Helping | pre-treatment, immediately post-treatment, 6-month follow-up, 12-month follow-up
  Parents and adolescents will complete the Helping for Health Inventory (Harris et al., 2008), a 15-item scale that measures miscarried helping or negative social support. Respondents rate on a 5-point scale the frequency with which parents engage in certain behaviors or feel certain ways pertaining to their child's health.

CONTACTS AND LOCATIONS:
Overall Officials: Tonya M. Palermo, Ph.D., Principal Investigator — University of Washington Medical School
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Result] Palermo TM, Law EF, Zhou C, Holley AL, Logan D, Tai G. Trajectories of change during a randomized controlled trial of internet-delivered psychological treatment for adolescent chronic pain: how does change in pain and function relate? Pain. 2015 Apr;156(4):626-634. doi: 10.1097/01.j.pain.0000460355.17246.6c. PMID 25775441
- [Derived] Law EF, Groenewald CB, Zhou C, Palermo TM. Effect on Health Care Costs for Adolescents Receiving Adjunctive Internet-Delivered Cognitive-Behavioral Therapy: Results of a Randomized Controlled Trial. J Pain. 2018 Aug;19(8):910-919. doi: 10.1016/j.jpain.2018.03.004. Epub 2018 Mar 22. PMID 29578090